CLINICAL TRIAL: NCT05759052
Title: Long-term Evaluation of Vincristine-induced Peripheral Neuropathy in Adult Survivors of a Multicenter Prospective Cohort of Childhood and Adolescent Leukemia (LEA Cohort): a Multicenter Cross-sectional Study
Brief Title: Vincristine-induced Peripheral Neuropathy in Adult Survivors of Childhood and Adolescent Leukemia
Acronym: CIPN-LEA
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC IR 2021 BALAYSSAC; 2022-A01758-35 (Other: ANSM)
Record Dates: First submitted 2023-02-13; First posted 2023-03-08 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: vincristine-induced peripheral neuropathy; pediatric leukemia; cancer survivor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of adult survivors having been treated by vincristine: Cohort of adult survivors having been treated by vincristine for a childhood leukemia
  Interventions: Behavioral: self-administered questionnaire

INTERVENTIONS:
Behavioral: self-administered questionnaire — Patients will answer to a self- administered questionnaire exploring chemotherapy-induced peripheral neuropathy and related comorbidities

SUMMARY:
Vincristine is a major anticancer agent in the management of hematological malignancies. One of the main side effects is chemotherapy-induced peripheral neuropathy (CIPN). CIPN is a characteristic side effect of neurotoxic anticancer drugs. CIPN associated with vincristine is typically characterized by distal and symmetrical sensory symptoms (dysesthesia and paresthesia). Motor and vegetative symptoms can also be found. The prevalence of CIPN associated with vincristine during treatment ranges from 12 to 100% in children (depending on the endpoint).

The aim of this cross-sectionnal study will be to explore the CIPN prevalence and severity in adult survivors of childhood leukemia and having been treated by vincristine.

DETAILED DESCRIPTION:
Adult survivors of chidlhood leukemia and having been treated by vincristine will be contacted from the French childhood cancer survivor study for leukaemia (LEA Cohort) in order to seek their participation agreement.

Thereafter patients will received a self-administered questionnaire exploring the chemotherapy-induced peripheral neuropathy and related comorbidities (pain, neuropathic pain, anxiety, depression, health-related quality of life, substance use, physical activity, deprivation). Oncological and sociodemographic characteristics of participants will be recorded.

ELIGIBILITY:
Inclusion Criteria:

- adult patient (> 18-year) who received a vincristine-based chemotherapy for hematological malignancy in childhood

Exclusion Criteria:

* Secondary cancer (leukemia and/or cancer)
* Active oncological pathology
* Current cancer treatment
* Adults protected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled from the French Childhood Cancer Survivor Study For Leukaemia (LEA Cohort), in each particiapting centers
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Sensitive chemotherapy-induced peripheral neuropathy | day 1
  Scores of the sensitive subscale of the QLQ-CIPN20 questionnaire (quality of life questionnaire - chemotherapy-induced peripheral neuropathy 20 questions) scores : 0 least - 100 worst

SECONDARY OUTCOMES:
Motor chemotherapy-induced peripheral neuropathy | day 1
  Scores of the motor subscale of the QLQ-CIPN20 questionnaire (quality of life questionnaire - chemotherapy-induced peripheral neuropathy 20 questions) scores : 0 least - 100 worst
Pain severity | day 1
  Scores of pain severirty assessed with a visual analogic scale scores : 0 no pain - 10 maximal pain
Neuropathic pain | day 1
  Scores of the DN4 interview questionnaire (Douleur neuropathique 4 questions) Scores : 0 least - 7 worst Threshold for neuropathic pain : 3
Ongoing analgesic treatment | day 1
  Reporting of ongoing analgesic treatment declared by the patient
Anxiety severity | day 1
  Scores of the anxiety subscale of the HADS questionnaire (Hospital anxiety and depression scale) Anxiety scores: 0 least - 21 worst Normal scores: ≤7 Borderline or suggestive of possible anxiety: 8-10 Indicative of anxiety: ≥11
Depression severity | day 1
  Scores of the depression subscale of the HADS questionnaire (Hospital anxiety and depression scale) Depression scores: 0 least - 21 worst Normal scores: ≤7 Borderline or suggestive of possible depression: 8-10 Indicative of depression: ≥11
Health-related quality of life | day 1
  Scores of the SF36 questionnaire (short-form 36) for each item: 0 worst - 100 best
Physical activity and sedentarity | day 1
  GPAQ questionnaire (Global Physical Activity Questionnaire) Work-related physical activity (minutes) Leisure-related physical activity (minutes) Time spent sitting (minutes)
Deprivation | day 1
  Scores of the EPICES questionnaire (Evaluation de la Précarité et des Inégalités de santé dans les Centres d'Examens de Santé) Scores: 0 best - 100 worst
Use of legal and illegal psychoactive drugs | day 1
  Reporting of legal psychoactive drug use (alcohol, tobacco, e-cigarette, psychoactive medication, cannabidiol, and other), and illegal psychoactive drug use (cannabis, and other)
Oncological characteristics | day 1
  Type of hematological malignancy and date of diagnosis ; Chemotherapy received: vincristine (date of last course and cumulative dose), anthracyclines (cumulative dose) ; Radiation therapy received: central nervous system irradiation and total dose, total body irradiation and total dose ; Hematopoietic stem cell (HSC) transplant: autograft or allograft, and date of transplant(s) ; Relapse (date)
Oncological characteristics | day 1
  Type of hematological malignancy, date of diagnosis, and relapse (date)
Anticancer drugs received | day 1
  vincristine (date of last course and cumulative dose), and anthracyclines (cumulative dose)
Radiation therapy received | day 1
  Central nervous system irradiation (total dose), total body irradiation (total dose)
Hematopoietic stem cell transplant | day 1
  Autograft or allograft, and date of transplant(s)
Sociodemographic characteristics | day 1
  Age at the time of the response to the study questionnaire ; Age at diagnosis of hematological malignancy ; Gender ; Weight, height, body surface area, weight-for-age and sex-percentile at diagnosis ; Weight, height and BMI at time of response ; Intercurrent pathology at time of response ; socio-professional group

CONTACTS AND LOCATIONS:
Overall Officials: David Balayssac, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France